CLINICAL TRIAL: NCT02855047
Title: The Prognostic Value of PGF and sFlt1 Variations Induced by the First Low-molecular-weight-heparin Injections in Women With Obstetrical Antiphospholipids Antibody Syndrome Starting a New Pregnancy and Following Treatment in Accordance With International Recommendations
Acronym: NOH-ANGIO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/JCG-02
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2016-07

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to evaluate plasmatic concentrations of free PGF and sFlt1 for blood samples taken before a first low-molecular-weight-heparin injection and also for blood samples taken on the 4th day of injections (the latter correspond to the first systematic control of platelet counts) in women who have an obstetric antiphospholipid antibody syndrome and who are initiating a new pregnancy with recommended treatment. Our goal is to test the prognostic value of these data on the occurrence of:

* pregnancy loss categorized as embryonic loss (before 10 weeks gestation), fetal death (before 20 weeks gestation), stillbirths (from 20 weeks gestation to delivery), and neonatal death defined before reaching 28 days of age.
* ischemic placental pathology (pre-eclampsia, retro-placental hematoma, birth of a small-for-gestational-age infant)

ELIGIBILITY:
Inclusion Criteria:

* Three unexplained consecutive spontaneous abortions before the 10th week of gestation (the recurrent embryo loss subgroup) - OR -
* One unexplained death of a morphologically normal fetus (fetal loss) at or after the 10th week of gestation (fetal loss subgroup).
* Women in the APS subgroup: persistently positive for LA, and/or aCL and/or aBeta2GP1
* Women initiating a new pregnancy during the 18 month observational period after obstetric APS diagnosis

Exclusion Criteria:

* Any history of thrombotic events or any treatment given during previous pregnancies that might have modified the natural course of the condition
* Women whose pregnancy losses could be explained by infectious, metabolic, anatomic or hormonal factors, or associated with paternal or maternal chromosomal causes
* Seropositivity for HIV, hepatitis B or C
* Women with antithrombin, protein C, or protein S deficiency, and women with abnormal fibrinogen or with the JAK2 V617F mutation were further excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were selected via the regional NOHA (Nîmes Obstetricians and Hematologists - Antiphospholipid Syndrome study) network, which referred women with losses of spontaneous pregnancies to the Hematology Outpatient Department of the Nîmes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2005-07; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Presence/absence of at least one of the following: preeclampsia, abruptio placenta, or fetal growth restriction (< 10th percentile) | 19 weeks gestation
  The primary endpoint was a composite outcome that included any of the following events occurring after 19 completed weeks during the observed pregnancy: preeclampsia, abruptio placenta, or fetal growth restriction (< 10th percentile), summarized as the so-called placenta-mediated complications PMCs.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Gris, MD, PhD, Study Director — Centre Hospitalier Universitiare de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémea, Nîmes, France

REFERENCES:
- [Result] Cochery-Nouvellon E, Mercier E, Bouvier S, Balducchi JP, Quere I, Perez-Martin A, Mousty E, Letouzey V, Gris JC. Obstetric antiphospholipid syndrome: early variations of angiogenic factors are associated with adverse outcomes. Haematologica. 2017 May;102(5):835-842. doi: 10.3324/haematol.2016.155184. Epub 2017 Jan 25. PMID 28126966